CLINICAL TRIAL: NCT03970408
Title: Effect of Neck Movements on Median Nerve Longitudinal Excursion During Neurodynamic Mobilization in Patients With Carpal Tunnel Syndrome
Brief Title: Median Nerve Excursion During Neurodynamic Mobilization
Status: Completed | Type: Observational
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Associate professor of Orthopedic Physical Therapy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: HMahmoud
Record Dates: First submitted 2019-05-25; First posted 2019-05-31 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-07

CONDITIONS: CTS
Keywords: Median nerve,; Carpal tunnel syndrome; Neurodynamic mobilization
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carpal tunnel syndrome: Patients with CTS who fulfill the following eligibility criteria:
  Inclusion criteria
  * Females and male patients referred with a CTS diagnosis confirmed by nerve conduction studies and positive Tinel and Phalen tests.
  * Age ranging from 30-50 years old.
  * The selected patient will be able to tolerate the entire standard neurodynamic technique.
  Exclusion criteria
  * Symptoms referred to the neck.
  * Sever CTS
  * More than 10% limitation of neck flexion, rotation, and side bending ranges.
  * History of disease, trauma, or surgery to neck, thorax, or upper limbs.
  * Presence of peripheral neuropathy or cervical radiculopathy.
  * History of systemic disease associated with neuropathies such as diabetes mellitus, connective tissue diseases, thyroid disease, or obesity.
  Interventions: Procedure: MNT1
- Healthy control: Asymptomatic healthy age-matched control with no symptoms or history of upper quadrant disease, dysfunction, trauma or surgery.
  Interventions: Procedure: MNT1

INTERVENTIONS:
Procedure: MNT1 — Participants will in supine. Arm will be position in standard MNT1. Shoulder, elbow, wrist and fingers will be maintained in the required position using a costumed splint throughout all testing.
  All movements will be limited to the range where pain or other symptoms are not provoked. Passive neck flexion and rotation will be added to MNT1 and will be applied as tensioning movements at level 3. All movements will be repeated three times and an average will be calculated. Myrin goniometer will be used to assess neck flexion and rotation. The movements order will be randomized using excel random generation function. Movements will be done by a single trained therapist. The end position will be held up to 10 seconds until median nerve excursion is recorded by US. For US capturing, the transducer will be positioned perpendicularly and aligned longitudinally with the median nerve at the wrist. Assessor will be blinded to participants grouping.
  Other Names: Neurodynamic tension test

SUMMARY:
This study will compare changes in longitudinal median nerve excursion when neck flexion and ipsilateral rotation are added to the standard Median neurodynamic test1 (MNT1) position in patients with carpal tunnel syndrome (CTS) and normal controls.

DETAILED DESCRIPTION:
Median nerve excursion will be assessed by ultrasonography during three positions: standard MNT1, neck flexion with MNT1, and ipsilateral rotation combined with MNT1. Both arms will be tested.

Arm will be held in abduction to 90° - 110° and external rotation to 90°, forearm supination, elbow extension and wrist and fingers extension using a custom made splint.

The standard MNT1 includes neck contralateral side flexion. Then, the researcher will move the neck passively into rotation and flexion. Passive range limit will be determined prior to testing using a goniometer and passive end feel. Movement order will be randomized using an excel random function.

Every position will be tested three times. A single researcher will do all movements passively. Nerve excursion will be measured in real time by the same ultrasonographer who is blinded to patients grouping.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate CTS.
* Must be able to tolerate the entire standard MNT1 position.

Exclusion Criteria:

* Severe CTS.
* Symptoms referred to the neck.
* Limited neck flexion, rotation, and side bending ranges (>10%).
* History of upper quadrant trauma, dysfunction or surgery.
* History of peripheral neuropathy or cervical radiculopathy.
* History of systemic disease associated with neuropathies such as diabetes mellitus, connective tissue diseases, thyroid disease, or obesity.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be selected from primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in longitudinal median nerve excursion with neck flexion | One day
  Changes in median nerve excursion, as measured by ultrasonography, when the neck is moved toward flexion combined with the standard MNT1
Changes in longitudinal median nerve excursion with ipsilateral neck rotation | One day
  Changes in median nerve excursion changes, as measured by ultrasonography, when the neck is moved in ipsilateral rotation combined with the standard MNT1

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, Phd, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Ain Shamas University, Cairo
  - Cairo University Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ballestero-Perez R, Plaza-Manzano G, Urraca-Gesto A, Romo-Romo F, Atin-Arratibel MLA, Pecos-Martin D, Gallego-Izquierdo T, Romero-Franco N. Effectiveness of Nerve Gliding Exercises on Carpal Tunnel Syndrome: A Systematic Review. J Manipulative Physiol Ther. 2017 Jan;40(1):50-59. doi: 10.1016/j.jmpt.2016.10.004. Epub 2016 Nov 11. PMID 27842937
- [Background] Balogun, J. a, & Abereoje, O. K. (1989). Inter- and lntratester Reliability of Measuring Neck Motions with Tape Measure and Myrin Gravity reference goniometer. Orthopaedic & Sports Physical Therapy, 10(7), 248-253.
- [Background] Bay BK, Sharkey NA, Szabo RM. Displacement and strain of the median nerve at the wrist. J Hand Surg Am. 1997 Jul;22(4):621-7. doi: 10.1016/S0363-5023(97)80118-9. PMID 9260616
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, Vincent KR, George SZ. A randomized sham-controlled trial of a neurodynamic technique in the treatment of carpal tunnel syndrome. J Orthop Sports Phys Ther. 2009 Oct;39(10):709-23. doi: 10.2519/jospt.2009.3117. PMID 19801812
- [Background] Botte MJ, von Schroeder HP, Abrams RA, Gellman H. Recurrent carpal tunnel syndrome. Hand Clin. 1996 Nov;12(4):731-43. PMID 8953292
- [Background] Boudier-Reveret M, Gilbert KK, Allegue DR, Moussadyk M, Brismee JM, Sizer PS Jr, Feipel V, Dugailly PM, Sobczak S. Effect of neurodynamic mobilization on fluid dispersion in median nerve at the level of the carpal tunnel: A cadaveric study. Musculoskelet Sci Pract. 2017 Oct;31:45-51. doi: 10.1016/j.msksp.2017.07.004. Epub 2017 Jul 17. PMID 28734168
- [Background] Brochwicz P, von Piekartz H, Zalpour C. Sonography assessment of the median nerve during cervical lateral glide and lateral flexion. Is there a difference in neurodynamics of asymptomatic people? Man Ther. 2013 Jun;18(3):216-9. doi: 10.1016/j.math.2012.10.001. Epub 2013 Jan 11. PMID 23317635
- [Background] Bueno-Gracia E, Ruiz-de-Escudero-Zapico A, Malo-Urries M, Shacklock M, Estebanez-de-Miguel E, Fanlo-Mazas P, Caudevilla-Polo S, Jimenez-Del-Barrio S. Dimensional changes of the carpal tunnel and the median nerve during manual mobilization of the carpal bones. Musculoskelet Sci Pract. 2018 Aug;36:12-16. doi: 10.1016/j.msksp.2018.04.002. Epub 2018 Apr 4. PMID 29635191
- [Background] Butler, D. S., & Jones, M. A. (1991). Mobilization of the Nervous System. In D. S. Butler & M. A. Jones (Eds.), clinical resoning (1st ed., pp. 91-105). Australia: Elsevier Health Sciences.
- [Background] Coppieters MW, Butler DS. Do 'sliders' slide and 'tensioners' tension? An analysis of neurodynamic techniques and considerations regarding their application. Man Ther. 2008 Jun;13(3):213-21. doi: 10.1016/j.math.2006.12.008. Epub 2007 Mar 30. PMID 17398140
- [Background] Coppieters MW, Hough AD, Dilley A. Different nerve-gliding exercises induce different magnitudes of median nerve longitudinal excursion: an in vivo study using dynamic ultrasound imaging. J Orthop Sports Phys Ther. 2009 Mar;39(3):164-71. doi: 10.2519/jospt.2009.2913. PMID 19252262
- [Background] De-la-Llave-Rincon AI, Ortega-Santiago R, Ambite-Quesada S, Gil-Crujera A, Puentedura EJ, Valenza MC, Fernandez-de-las-Penas C. Response of pain intensity to soft tissue mobilization and neurodynamic technique: a series of 18 patients with chronic carpal tunnel syndrome. J Manipulative Physiol Ther. 2012 Jul;35(6):420-7. doi: 10.1016/j.jmpt.2012.06.002. Epub 2012 Jul 31. PMID 22858234
- [Background] Dilley A, Lynn B, Greening J, DeLeon N. Quantitative in vivo studies of median nerve sliding in response to wrist, elbow, shoulder and neck movements. Clin Biomech (Bristol). 2003 Dec;18(10):899-907. doi: 10.1016/s0268-0033(03)00176-1. PMID 14580833
- [Background] Duncan, S. F. M., & Kakinoki Ryosuke. (2017). Carpal Tunnel Syndrome and Related Median Neuropathies. In M. E. Cooke & S. F. M. Duncan (Eds.), Challenges and Complications. (1st ed., pp. 7-11). USA: Springer.
- [Background] Echigo A, Aoki M, Ishiai S, Yamaguchi M, Nakamura M, Sawada Y. The excursion of the median nerve during nerve gliding exercise: an observation with high-resolution ultrasonography. J Hand Ther. 2008 Jul-Sep;21(3):221-7; quiz 228. doi: 10.1197/j.jht.2007.11.001. PMID 18652966
- [Background] Ellis R, Blyth R, Arnold N, Miner-Williams W. Is there a relationship between impaired median nerve excursion and carpal tunnel syndrome? A systematic review. J Hand Ther. 2017 Jan-Mar;30(1):3-12. doi: 10.1016/j.jht.2016.09.002. Epub 2016 Sep 28. PMID 27692791
- [Background] Ferry S, Pritchard T, Keenan J, Croft P, Silman AJ. Estimating the prevalence of delayed median nerve conduction in the general population. Br J Rheumatol. 1998 Jun;37(6):630-5. doi: 10.1093/rheumatology/37.6.630. PMID 9667616
- [Background] Foley M, Silverstein B, Polissar N. The economic burden of carpal tunnel syndrome: long-term earnings of CTS claimants in Washington State. Am J Ind Med. 2007 Mar;50(3):155-72. doi: 10.1002/ajim.20430. PMID 17216630
- [Background] Ginanneschi F, Cioncoloni D, Bigliazzi J, Bonifazi M, Lore C, Rossi A. Sensory axons excitability changes in carpal tunnel syndrome after neural mobilization. Neurol Sci. 2015 Sep;36(9):1611-5. doi: 10.1007/s10072-015-2218-x. Epub 2015 Apr 21. PMID 25896622
- [Background] Gonzalezsuarez, C., Nathleendizon, J., Cua, R., Cabungcalfidel, B., Dones, V., Lesniewski, P., & Thomas, J. C. (2016). Determination of the longitudinal median nerve mobility in different neurodynamic techniques. Hand Therapy, 21(1), 16-24.
- [Background] Heebner ML, Roddey TS. The effects of neural mobilization in addition to standard care in persons with carpal tunnel syndrome from a community hospital. J Hand Ther. 2008 Jul-Sep;21(3):229-40; quiz 241. doi: 10.1197/j.jht.2007.12.001. PMID 18652967
- [Background] Hough AD, Moore AP, Jones MP. Reduced longitudinal excursion of the median nerve in carpal tunnel syndrome. Arch Phys Med Rehabil. 2007 May;88(5):569-76. doi: 10.1016/j.apmr.2007.02.015. PMID 17466724
- [Background] Hsieh, Y. H., Shih, J. T., Lee, H. M., & Ho, Y. J. (2010). Ultrasonography of median nerve mobility in the diagnosis of carpal tunnel syndrome. Formosan Journal of Musculoskeletal Disorders, 1(1), 16-19.
- [Background] Kantarci F, Ustabasioglu FE, Delil S, Olgun DC, Korkmazer B, Dikici AS, Tutar O, Nalbantoglu M, Uzun N, Mihmanli I. Median nerve stiffness measurement by shear wave elastography: a potential sonographic method in the diagnosis of carpal tunnel syndrome. Eur Radiol. 2014 Feb;24(2):434-40. doi: 10.1007/s00330-013-3023-7. Epub 2013 Sep 25. PMID 24220753
- [Background] Korstanje JW, Scheltens-De Boer M, Blok JH, Amadio PC, Hovius SE, Stam HJ, Selles RW. Ultrasonographic assessment of longitudinal median nerve and hand flexor tendon dynamics in carpal tunnel syndrome. Muscle Nerve. 2012 May;45(5):721-9. doi: 10.1002/mus.23246. PMID 22499100
- [Background] Kostopoulos, D. (2004). Treatment of carpal tunnel syndrome : a review of the non-surgical approaches with emphasis in neural mobilization. Journal of Bodywork and Movement Therapies, 8(1), 2-8.
- [Background] Lopes MM, Lawson W, Scott T, Keir PJ. Tendon and nerve excursion in the carpal tunnel in healthy and CTD wrists. Clin Biomech (Bristol). 2011 Nov;26(9):930-6. doi: 10.1016/j.clinbiomech.2011.03.014. Epub 2011 May 8. PMID 21550703
- [Background] Luchetti, R., & Amadio, P. (2007). Normal anatomy and variations of the median nerve in the carpal tunnel. In H. M. Schmidt (Ed.), Carpal Tunnel Syndrome (pp. 13-20). Berlin Heidelberg: Springer.
- [Background] McLellan DL, Swash M. Longitudinal sliding of the median nerve during movements of the upper limb. J Neurol Neurosurg Psychiatry. 1976 Jun;39(6):566-70. doi: 10.1136/jnnp.39.6.566. PMID 950567
- [Background] Meng S, Reissig LF, Beikircher R, Tzou CH, Grisold W, Weninger WJ. Longitudinal Gliding of the Median Nerve in the Carpal Tunnel: Ultrasound Cadaveric Evaluation of Conventional and Novel Concepts of Nerve Mobilization. Arch Phys Med Rehabil. 2015 Dec;96(12):2207-13. doi: 10.1016/j.apmr.2015.08.415. Epub 2015 Aug 24. PMID 26315068
- [Background] Mohamed, F., Hassan, A., Abdel-Magied, R., & Wageh, R. (2016). Manual therapy intervention in the treatment of patients with carpal tunnel syndrome: median nerve mobilization versus medical treatment. Egyptian Rheumatology and Rehabilitation, 43(1), 27-34.
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240
- [Background] Paquette P, Lamontagne M, Higgins J, Gagnon DH. Repeatability and Minimal Detectable Change in Longitudinal Median Nerve Excursion Measures During Upper Limb Neurodynamic Techniques in a Mixed Population: A Pilot Study Using Musculoskeletal Ultrasound Imaging. Ultrasound Med Biol. 2015 Jul;41(7):2082-6. doi: 10.1016/j.ultrasmedbio.2015.03.015. Epub 2015 Apr 11. PMID 25868536
- [Background] Polykandriotis E, Premm W, Horch RE. Carpal tunnel syndrome in young adults--an ultrasonographic and neurophysiological study. Minim Invasive Neurosurg. 2007 Dec;50(6):328-34. doi: 10.1055/s-2007-993163. PMID 18210354
- [Background] Schmid AB, Elliott JM, Strudwick MW, Little M, Coppieters MW. Effect of splinting and exercise on intraneural edema of the median nerve in carpal tunnel syndrome--an MRI study to reveal therapeutic mechanisms. J Orthop Res. 2012 Aug;30(8):1343-50. doi: 10.1002/jor.22064. Epub 2012 Jan 9. PMID 22231571
- [Background] Shacklock, M. (2005). Clinical Neurodynamics: In A new system of musculoskeletal treatment (1st ed., pp. 22-121). Australia: Elsevier Health Sciences.
- [Background] Silva A, Manso A, Andrade R, Domingues V, Brandao MP, Silva AG. Quantitative in vivo longitudinal nerve excursion and strain in response to joint movement: A systematic literature review. Clin Biomech (Bristol). 2014 Sep;29(8):839-47. doi: 10.1016/j.clinbiomech.2014.07.006. Epub 2014 Aug 10. PMID 25168082
- [Background] Suk JI, Walker FO, Cartwright MS. Ultrasonography of peripheral nerves. Curr Neurol Neurosci Rep. 2013 Feb;13(2):328. doi: 10.1007/s11910-012-0328-x. PMID 23314937
- [Background] Tal-Akabi A, Rushton A. An investigation to compare the effectiveness of carpal bone mobilisation and neurodynamic mobilisation as methods of treatment for carpal tunnel syndrome. Man Ther. 2000 Nov;5(4):214-22. doi: 10.1054/math.2000.0355. PMID 11052900
- [Background] Tat J, Wilson KE, Keir PJ. Pathological changes in the subsynovial connective tissue increase with self-reported carpal tunnel syndrome symptoms. Clin Biomech (Bristol). 2015 May;30(4):360-5. doi: 10.1016/j.clinbiomech.2015.02.015. Epub 2015 Mar 2. PMID 25753696
- [Background] Valls-Sole J, Alvarez R, Nunez M. Limited longitudinal sliding of the median nerve in patients with carpal tunnel syndrome. Muscle Nerve. 1995 Jul;18(7):761-7. doi: 10.1002/mus.880180713. PMID 7783766
- [Background] van Doesburg MH, Henderson J, Yoshii Y, Mink van der Molen AB, Cha SS, An KN, Amadio PC. Median nerve deformation in differential finger motions: ultrasonographic comparison of carpal tunnel syndrome patients and healthy controls. J Orthop Res. 2012 Apr;30(4):643-8. doi: 10.1002/jor.21562. Epub 2011 Sep 27. PMID 21953849
- [Background] van Doesburg MH, Mink van der Molen A, Henderson J, Cha SS, An KN, Amadio PC. Sonographic measurements of subsynovial connective tissue thickness in patients with carpal tunnel syndrome. J Ultrasound Med. 2012 Jan;31(1):31-6. doi: 10.7863/jum.2012.31.1.31. PMID 22215766
- [Background] Wang Y, Zhao C, Passe SM, Filius A, Thoreson AR, An KN, Amadio PC. Transverse ultrasound assessment of median nerve deformation and displacement in the human carpal tunnel during wrist movements. Ultrasound Med Biol. 2014 Jan;40(1):53-61. doi: 10.1016/j.ultrasmedbio.2013.09.009. Epub 2013 Nov 7. PMID 24210862
- [Background] Wolny T, Linek P. Neurodynamic Techniques Versus "Sham" Therapy in the Treatment of Carpal Tunnel Syndrome: A Randomized Placebo-Controlled Trial. Arch Phys Med Rehabil. 2018 May;99(5):843-854. doi: 10.1016/j.apmr.2017.12.005. Epub 2018 Jan 4. PMID 29307812
- [Background] Wolny T, Saulicz E, Linek P, Mysliwiec A, Saulicz M. Effect of manual therapy and neurodynamic techniques vs ultrasound and laser on 2PD in patients with CTS: A randomized controlled trial. J Hand Ther. 2016 Jul-Sep;29(3):235-45. doi: 10.1016/j.jht.2016.03.006. Epub 2016 Apr 16. PMID 27094495
- [Background] Wolny T, Saulicz E, Linek P, Shacklock M, Mysliwiec A. Efficacy of Manual Therapy Including Neurodynamic Techniques for the Treatment of Carpal Tunnel Syndrome: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2017 May;40(4):263-272. doi: 10.1016/j.jmpt.2017.02.004. Epub 2017 Apr 8. PMID 28395984